CLINICAL TRIAL: NCT07363291
Title: Standardized Implementation and Quality Assessment System for Confocal Enteroscopy
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Huashan Hospital (Other); Renji Hospital Anhui Hospital (Unknown); Ruijin Hospital (Other); Kashgar Second People's Hospital (Unknown); Ningbo Hangzhou Bay Hospital (Unknown)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Other Study IDs: KY2024-200-B
Record Dates: First submitted 2025-10-01; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Confocal Enteroscopy; Quality Assessment System; Standardized Implementation
Keywords: Confocal Enteroscopy; Standardized Implementation; Quality Assessment System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Confocal Enteroscopy group: Record the performance under CLE
- Conventional enteroscopy group: Record the performance under Enteroscopy

SUMMARY:
Confocal technology, hailed as "optical biopsy," enables real-time cellular-level histological examination of mucosal surfaces. Its integration with double-balloon enteroscopy significantly enhances the clinical feasibility of targeted biopsy, early diagnosis, and endoscopic staging for small bowel diseases such as inflammatory bowel disease. Currently, confocal endoscopy is primarily applied to upper and lower gastrointestinal tract diseases, leaving small bowel pathologies largely unexplored. Consequently, establishing a diagnostic framework for small bowel tumors and non-neoplastic lesions using confocal enteroscopy, alongside developing quality assessment standards for its operational procedures, is of paramount importance.

DETAILED DESCRIPTION:
This project intends to establish a multi-center cohort comprising 200 confocal small-bowel endoscopy cases plus 400 gastrointestinal control cases, equally split into two arms: an exploratory arm and a validation arm. Controls will be selected according to the research objective: for neoplastic lesions, normal-appearing small bowel, colonic adenomas, and early gastric adenocarcinoma; for non-neoplastic lesions, normal-appearing small bowel, colonic segments involved by IBD, and gastric segments involved by IBD.

Main inclusion: patients with suspected small-bowel disease who require endoscopy for lesion characterization, including but not limited to clinically suspected active or quiescent small-bowel Crohn's disease with or without complications, unclassified IBD such as CMUSE, hereditary small-bowel neoplastic syndromes (e.g. Peutz-Jeghers), and small-bowel lymphomas that need endoscopy plus histology.

During single- or double-balloon enteroscopy, areas endoscopically suspected and adjacent normal mucosa will be examined with confocal laser endomicroscopy (CLE). Conventional enteroscopic and CLE findings will be summarized; CLE variables will include, but are not limited to, mucosal-barrier assessment (epithelial gap score, cell-shedding score, Watson score), inflammatory activity based on crypt architecture, ENHANCE mucosal-healing score, and will be augmented by AI image-recognition systems (Yingnuo™ & Xiaohua-Tanying™).

Using the exploratory arm, parameters that show statistically significant contribution to diagnosis by integrating endoscopic and comprehensive clinical diagnosis will be identified to build a new confocal enteroscopy-based model for small-bowel IBD, which will then be tested in the validation arm for sensitivity, specificity, AUC, etc. The auxiliary role of AI in lesion recognition will also be evaluated.

In parallel, quality-control (QC) indicators will be developed from the clinical-use cohort. Key indicators include: procedural-success rate (proportion of completed confocal enteroscopies), diagnostic accuracy (concordance with pathology or gold standard, including AI-induced drift), adverse-event rate, and image-quality score.

Contributions to QC of the entire workflow-pre-procedure (scope model, CLE mode setting, patient risk/anesthesia assessment, demographics), intra-procedure (insertion/withdrawal time, time to lesion, scope posture, completeness of CLE parameters, bowel preparation), and post-procedure (specimen handling, recovery, observation time, prophylactic antibiotics)-will be quantified by logistic regression to identify high-impact factors and build a scientific QC system. This system will be applied to the validation arm for feasibility and accuracy, and regular internal audits will be conducted for continuous improvement.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years and scheduled to undergo small-bowel endoscopy.
* Able to provide written informed consent and willing to participate in the study.
* Certified gastroenterologists with an intermediate (or higher) professional title.

Have completed formal training and passed competency assessments in gastroscopy, colonoscopy, and small-bowel endoscopy.

-Willing to participate and able to provide written informed consent.

Exclusion Criteria:

* Poor general condition, severe hepatic or renal insufficiency, or inability to tolerate complete endoscopic examination.
* Known hypersensitivity to any study-related agents (fluorescein sodium, polyethylene glycol, lidocaine mucilage).
* Currently enrolled in another clinical trial.
* Never perform endoscopic procedures.
* Endoscopic procedure or image-reading volume < 100 cases in the past 2 years.
* Medical license revoked or currently suspended for any reason.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Aged 18-70 years and scheduled to undergo small-bowel endoscopy.
  * Able to provide written informed consent and willing to participate in the study.
  * Certified gastroenterologists with an intermediate (or higher) professional title.
  Have completed formal training and passed competency assessments in gastroscopy, colonoscopy, and small-bowel endoscopy.
  -Willing to participate and able to provide written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
procedural success rate | 14 days
  the proportion of examinations in which confocal enteroscopy was successfully completed

SECONDARY OUTCOMES:
diagnostic accuracy | 14 days
  the proportion of clinical findings that are consistent with pathology or other gold-standard diagnoses, and the impact of AI-induced bias on this concordance
complication rate | 14 days
  the number of cases in which complications occur after the examination

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Renji Hospital Anhui Hospital, Hefei, Anhui
  - Ningbo Hangzhou Bay Hospital, Ningbo, Zhejiang
  - Kashgar Second People's Hospital, Kashgar
  - Huashan Hospital, Fudan University, Shanghai
  - Renji Hospital, Shanghai
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No